CLINICAL TRIAL: NCT01399190
Title: An Open Label Study of the Effect of First Line Treatment With Bevacizumab in Combination With Capecitabine and Oxaliplatin on Progression-free Survival in Patients With Metastatic Cancer of the Colon and Rectum
Brief Title: An Observational Study of Avastin (Bevacizumab) in Combination With Xeloda (Capecitabine) And Oxaliplatin in Patients With Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25523
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Bevacizumab: Participants will receive bevacizumab in combination with capecitabine and oxaliplatin.
  Interventions: Biological: Bevacizumab; Biological: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Bevacizumab — Bevacizumab administered according to prescribing information and normal clinical practice.
  Other Names: Avastin®
Biological: Capecitabine — Capecitabine administered according to prescribing information and normal clinical practice.
  Other Names: Xeloda®
Drug: Oxaliplatin — Capecitabine administered according to prescribing information and normal clinical practice.
  Other Names: Eloxatin™

SUMMARY:
This prospective observational study will evaluate the efficacy and safety of bevacizumab in combination with capecitabine and oxaliplatin as first-line treatment in participants with colorectal cancer. Data will be collected from each participant until disease progression occurs (for up to 30 months).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Metastatic colorectal cancer
* Treatment in accordance with current Summary of Product Characteristics and local guidelines

Exclusion Criteria:

* Contraindications according to current Summary of Product Characteristics and local guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with colorectal cancer on first-line treatment with bevacizumab in combination with capecitabine and oxaliplatin.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Slovakia (8):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Martin
  - Nitra
  - Poprad
  - Prešov
  - Ružomberok

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Participants received bevacizumab in combination with capecitabine and oxaliplatin according to prescribing information and normal clinical practice.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 68
Included in Final Analysis | 63
Evaluable for Primary Endpoint Analysis | 60
Completed | 48
Not Completed | 20
Not completed — Not Eligible for Final Analysis | 5
Not completed — Adverse Event | 8
Not completed — Participant's Request | 5
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Includes enrolled participants eligible for inclusion in the final analysis.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.08 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the interval between the day of first treatment and the first documentation of disease progression or death and was assessed by the investigators according to modified Response Evaluation Criteria in Solid Tumors (RECIST). Disease progression was defined as an increase in sum of lesions size by more than 20% or new lesions.
Time Frame: From randomization to progression or death during the study (up to approximately 30 months)
Population: Includes enrolled participants who were evaluable for the primary endpoint analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 60
months | 7.000 [5.577 to 8.423]

2. Secondary Outcome: Response Rate (Tumor Assessments According to RECIST)
Description: Response to treatment (Response Rate) was defined as the percentage of participants with a complete remission (CR) or partial remission (PR), and was assessed by the investigators according to modified RECIST criteria. CR was defined as disappearance of all lesions. PR was defined as a decrease in sum of lesions size by more than 30%. Response Rate = CR +PR
Time Frame: Up to approximately 30 months
Population: Includes enrolled participants who were evaluable for the primary endpoint analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 60
percentage of participants
  Response Rate | 48.4
  Complete remission | 6.7
  Partial remission | 41.7

3. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to approximately 30 months
Population: Includes enrolled participants eligible for inclusion in the final analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 63
percentage of participants | 74.6

ADVERSE EVENTS:
Time Frame: Up to approximately 30 months
Description: Includes enrolled participants eligible for inclusion in the final analysis.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 2/63
Other Adverse Events (participants affected / at risk) | 39/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=63)
Hypertensive crisis (Vascular disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=63)
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Allergic reaction (Immune system disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 23
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.